CLINICAL TRIAL: NCT04025216
Title: A Phase 1 Open-Label, Multi-Center First in Human Study of TnMUC1-Targeted Genetically-Modified Chimeric Antigen Receptor T Cells in Patients With Advanced TnMUC1-Positive Solid Tumors and Multiple Myeloma
Brief Title: A Study of CART-TnMUC1 in Patients With TnMUC1-Positive Advanced Cancers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The sponsor finds the risk/benefit analysis unfavorable and has terminated the study.
Sponsor: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CART-TnMUC1-01
Record Dates: First submitted 2019-07-12; First posted 2019-07-18 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2023-04

CONDITIONS: Non-Small Cell Lung Cancer; Ovarian Cancer; Fallopian Tube Cancer; Triple Negative Breast Cancer; Multiple Myeloma; Pancreatic Ductal Adenocarcinoma
Keywords: Chimeric Antigen Receptor (CAR); T-cells; TnMUC1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms; Fallopian Tube Neoplasms; Triple Negative Breast Neoplasms; Multiple Myeloma | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Intervention Model Description: Parallel arms with sequential dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Arm1: Solid Tumors (Experimental): Intravenous CART-TnMUC1 cells for patients with TnMUC1+ treatment-resistant ovarian cancer (including cancers of the fallopian tube), pancreatic ductal adenocarcinoma, hormone receptor (HR)-negative and human epidermal growth factor receptor 2 (HER2)-negative (triple negative) breast cancer and non-small cell lung cancer
  Interventions: Biological: CART-TnMUC1; Drug: Cyclophosphamide; Drug: Fludarabine
- Dose Escalation Arm 2: Multiple Myeloma (Experimental): Intravenous CART-TnMUC1 cells for patients with TnMUC1+ relapsed/refractory multiple myeloma
  Interventions: Biological: CART-TnMUC1; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: CART-TnMUC1 — Single intravenous administration of genetically modified autologous T cells engineered to express a TnMUC1-Targeted Genetically-Modified Chimeric Antigen (CAR)
Drug: Cyclophosphamide — Patients will receive cyclophosphamide and fludarabine lymphodepletion chemotherapy followed by the investigational product, CART-TnMUC1
Drug: Fludarabine — Patients will receive cyclophosphamide and fludarabine lymphodepletion chemotherapy followed by the investigational product, CART-TnMUC1

SUMMARY:
Multi-center, open-label, first in human Phase 1 study of the safety, tolerability, feasibility, and preliminary efficacy of the administration of genetically modified autologous T cells (CART-TnMUC1 cells) engineered to express a chimeric antigen receptor (CAR) capable of recognizing the tumor antigen, TnMUC1 and activating the T cell (CART- TnMUC1 cells).

DETAILED DESCRIPTION:
The Dose Escalation phase of the study is designed to identify the dose and regimen of CART-TnMUC1 cells that can be safely administered intravenously following the lymphodepletion (LD) regimen to patients with (1) advanced TnMUC1+ solid tumors (triple negative breast cancer, epithelial ovarian cancer, pancreatic cancer, and non-small cell lung cancer) and (2) advanced TnMUC1+ multiple myeloma in a parallel two-arm dose escalation study. The Dose Escalation phase is anticipated to enroll approximately 40 patients.

The Expansion phase of the study is designed to assess the preliminary efficacy of CART-TnMUC1 cells administered intravenously to patients with TnMUC1+ solid tumors. The Expansion phase is anticipated to enroll approximately 72 patients (18 patients per each tumor indication).

ELIGIBILITY:
Key Inclusion Criteria:

* Confirmed diagnosis of metastatic treatment-resistant ovarian cancer (including cancers of the fallopian tube), pancreatic adenocarcinoma, hormone receptor (HR)-negative and HER2-negative (triple negative) breast cancer (TNBC) or non-small cell lung cancer (NSCLC), or relapsed/refractory multiple myeloma
* Eastern Cooperative Oncology Group (ECOG) score of 0 or 1
* Prior therapies as defined by tumor type:

  * Multiple myeloma: relapsed or refractory disease previously treated with or intolerant to at least three different lines of therapy that contained at least one of the following drug classes: proteasome inhibitor, an immune modulatory drug, alkylators, CD38 monoclonal antibody and glucocorticoids. Patients must be at least 90 days since autologous stem cell transplant
  * NSCLC: i.) Patients without driver mutations must have received standard therapy, including both checkpoint inhibition and platinum-based chemotherapy or be intolerant of these standard therapies ii.) Patients with driver mutations must have received or be intolerant to prior targeted therapy directed at the specific identified mutations in addition to the standard chemotherapy classes
  * Pancreatic adenocarcinoma: disease progression following at least one standard of care systemic chemotherapy for metastatic or unresectable disease or be intolerant of these standard therapies
  * TNBC: ER and/or PR < or =10%, HER2 negative and experienced disease progression following at least one prior systemic anti-cancer therapy regimen as part of their treatment for management of metastatic breast cancer or be intolerant to these standard therapies
  * Ovarian: platinum-resistant (progression of disease by either CA-125, clinical or radiographic assessment within 6 months of last platinum-based chemotherapy ) and must have received at least two prior lines of therapy for metastatic ovarian cancer, including at least one prior line of therapy including a platinum-containing regimen or be intolerant of these standard therapies
* Evaluable disease as defined by tumor type
* TnMUC1+ disease, determined by centrally tested TnMUC1 expression in a prior or archival tumor biopsy
* Toxicities from any previous therapy must have recovered to Grade 1 or baseline
* Estimated estimated glomerular filtration rate ≥ 60 m/min by Modification of Diet in Renal Disease criteria
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 2.5 x upper institutional limit of normal with the following exception: Patients with known hepatic metastases, AST or ALT ≤ 3 x upper institutional limit of normal
* Serum total bilirubin < 1.5 mg/dL with the following exception: patients with known Gilbert's disease, serum total bilirubin < 3 mg/dL
* Serum albumin ≥ 3.0 g/dL (solid tumor patients in Arm 1 and Phase 1a only, not applicable to patients with multiple myeloma)
* Left ventricular ejection fraction (LVEF) ≥ 50%. LVEF assessment must have been performed within 6 months of treatment start
* Hemoglobin ≥ 8 g/dL
* Absolute neutrophil count ≥ 1000/μL
* Platelet count ≥ 75,000/μL (for Multiple Myeloma patients with bone marrow plasma cells ≥ 50% of cellularity: ≥ 30,000/μL)
* Patients of reproductive potential agree to use approved contraceptive methods per protocol

Key Exclusion Criteria:

* Active invasive cancer other than the proposed cancers included in the study
* Current treatment with systemic high-dose corticosteroids (defined as a dose greater than the equivalent of prednisone 10 mg/day)
* Active autoimmune disease (including connective tissue disease, uveitis, sarcoidosis, inflammatory bowel disease or multiple sclerosis) or have a history of severe autoimmune disease requiring prolonged immunosuppressive therapy (any immunosuppressive therapy should have been stopped within 6 weeks prior to screening visit)
* Current human immunodeficiency virus (HIV), hepatitis C virus (HCV), hepatitis B virus (HBV) infections
* Other active or uncontrolled medical or psychiatric condition that would preclude participation in the opinion of the Sponsor or Principal Investigator
* Prior allogeneic stem cell transplant
* Active and untreated central nervous system (CNS) malignancy
* History of severe infusion reaction to monoclonal antibodies or biological therapies, or to study product excipients that would preclude the patient safely receiving CART-TnMUC1 cells
* Active or recent (within the past 6 months prior to apheresis) cardiovascular disease, defined as (1) New York Heart Association (NYHA) Class III or IV heart failure, (2) unstable angina or (3) a history of recent (within 6 months) myocardial infarction or sustained (> 30 second) ventricular tachyarrhythmias, or (4) cerebrovascular accident
* Have inadequate venous access for or contraindications for the apheresis procedure
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
Dose Escalation: Dose Identification of CART-TnMUC1 | Up to 2 years
  Incidence of Dose Limiting Toxicity (DLT) in solid tumors and multiple myeloma
Cohort Expansion: Objective Response in solid tumors | Up to 2 years
  Proportion of patients having a confirmed Complete Response (CR) or Partial Response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

SECONDARY OUTCOMES:
Safety of CART-TnMUC1 in solid tumors and multiple myeloma | Up to 2 years
  Percentage of patients experiencing adverse events (AEs), including serious and severe AEs overall, by dose level, and by severity Grade
Tolerability of CART-TnMUC1 in solid tumors and multiple myeloma | Up to 2 years
  Frequency of treatment emergent AEs, frequency of clinical changes from baseline in vital signs, changes in electrocardiogram, and hematology and chemistry laboratory shifts from baseline
Feasibility of CART-TnMUC1 in solid tumors and multiple myeloma | Up to 2 years
  Proportion of enrolled patients who did not receive CART-TnMUC1 cells
Preliminary anti-tumor efficacy of CART as assessed by Overall Survival (OS) in solid tumors and multiple myeloma | Up to 2 years
  OS as defined by the interval between CART-TnMUC1 cell infusion and date of death by any cause
Preliminary anti-tumor efficacy of CART as assessed by Progression Free Survival (PFS) in solid tumors | Up to 2 years
  PFS as defined by the interval between CART-TnMUC1 cell infusion and date of disease progression by RECIST v1.1 or death in solid tumors and by International Myeloma Working Group (IMWG) criteria in multiple myeloma
Preliminary anti-tumor efficacy of CART as assessed by Objective Response Rate (ORR) in solid tumors and multiple myeloma | Up to 2 years
  Proportion of patients having a confirmed CR or PR per RECIST v1.1 in solid tumors and IMWG criteria (PR, Very Good PR, CR, Stringent CR) in multiple myeloma
Preliminary anti-tumor efficacy of CART as assessed by Clinical Benefit Rate in solid tumors | Up to 2 years
  Proportion of patients having a confirmed CR, PR, or Stable Disease (SD) per RECIST v1.1
Preliminary anti-tumor efficacy of CART as assessed by Duration of Response (DOR) in solid tumors and multiple myeloma | Up to 2 years
  DOR as defined by the interval of first documented response until first documented disease progression or death in solid tumors and multiple myeloma
Preliminary anti-tumor efficacy of CART as assessed by Time to Response (TTR) in solid tumors and multiple myeloma | Up to 2 years
  Time to Response as defined by the interval between CART-TnMUC1 cell infusion and first documented CR or PR per RECIST v1.1 in solid tumors and IMWG criteria in multiple myeloma
Preliminary anti-tumor efficacy of CART as assessed by Time to Progression (TTP) in multiple myeloma | Up to 2 years
  Time to Progression as defined by the interval between CART-TnMUC1 cell infusion and first documented progression or death due to disease per RECIST v1.1 in solid tumors and IMWG criteria in multiple myeloma
Preliminary anti-tumor efficacy of CART as assessed by Minimal Residual Disease (MRD) in multiple myeloma | Up to 2 years
  Defined by MRD-negative rate per IMWG criteria
Peripheral expansion and persistence of CART-TnMUC1 cells in solid tumors and multiple myeloma | Up to 15 years
  Defined as quantitative polymerase chain reaction (qPCR) documenting loss of CART cells

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Mayo Clinic of Arizona, Phoenix, Arizona
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - Moffitt Cancer Center, Tampa, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Washington University School of Medicine, St Louis, Missouri
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No